CLINICAL TRIAL: NCT06139458
Title: Use of Cryocompression to Reduce Chemotherapy-induced Peripheral Neuropathy in Gynecologic Cancer: a Randomized Controlled Trial - COHORT 2
Brief Title: Cryocompression to Reduce Chemotherapy-induced Peripheral Neuropathy in Gynecologic Cancer - COHORT 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00106236_1
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Gynecologic Cancer; Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy (Experimental)
  Interventions: Behavioral: Cryotherapy
- Compression with Cryotherapy (Experimental)
  Interventions: Behavioral: Cryotherapy; Behavioral: Compression

INTERVENTIONS:
Behavioral: Cryotherapy — Participants will receive cryotherapy on both hands and feet
Behavioral: Compression — Participants will receive compression on both hands and feet
  Arms: Compression with Cryotherapy

SUMMARY:
The investigators aim to determine the effect of cryotherapy wraps plus compression therapy (henceforth referred to as cryocompression) versus cryotherapy wraps alone on the incidence and degree of chemotherapy-induced peripheral neuropathy in patients with gynecologic cancer using a noninferiority design. The investigators also aim to determine the effect of cryocompression versus cryotherapy on patient tolerability and patient and staff satisfaction.

DETAILED DESCRIPTION:
Participants will be randomized by patient to receive cryotherapy wraps plus compression therapy (cryocompression) versus cryotherapy wraps alone applied to the bilateral hands and feet. Participants will receive cryotherapy (+/- compression) for the duration of their taxane infusions. Participants will be asked to complete the FACT-NTX survey and a PNQ neuropathy surveys at each infusion visit to evaluate symptoms related to neuropathy. Participants will also complete a brief acceptability and tolerability survey at each visit. Lastly, a staff satisfaction survey will be administered at each visit as well. The investigators will test the hypothesis that the average final visit FACT-NTX11 scores in the cryotherapy group are noninferior to the cryocompression group with a noninferiority margin of 2.5 points. The investigators will routinely monitor for the following adverse events: frost bite, (unexpected) hospitalizations, and death.

ELIGIBILITY:
Inclusion Criteria:

* Gynecologic cancer diagnosis (ovarian, cervical, endometrial cancer; adenocarcinomas of likely primary gynecologic origin based on cytology or FNA in conjunction with radiologic impression will be eligible)
* Plan to receive at least 6 cycles of paclitaxel administered every 3 weeks at the Duke Cancer Center or Macon Pond or at the Carilion Clinic in Roanoke, VA. Patients receiving neoadjuvant chemotherapy with a plan for interval debulking will be eligible.
* ECOG (Eastern Cooperative Oncology Group) performance status of 0-1

Exclusion Criteria:

* Treated with prior neurotoxic chemotherapeutic agents
* Baseline diagnosis of peripheral neuropathy such as diabetic neuropathy, or conditions including but not limited to fibromyalgia, cryoglobulinemia and Raynaud's disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Assessment of Cancer Therapy (FACT) -Taxane [FACT-NTX] (patient reported assessment) over time | Up to two months after completion of chemotherapy, an average of 6 months
  The FACT-NTX is a patient self-reported 11-item questionnaire used for evaluating symptoms and concerns specifically associated with chemotherapy induced neuropathy. The total score ranges from 0-44, and a lower FACT-NTX score corresponds to worsening neuropathy. For both the FACT-NTX and the sensory subscale of the FACT-NTX, a significant decrease in the score is defined as a decrease exceeding 10% from baseline.

SECONDARY OUTCOMES:
Tolerability of cryocompression: scale | Up to two months after completion of chemotherapy, an average of 6 months
  Subjects will be asked to complete a cryocompression tolerability assessment after each chemotherapy session in which they will answer the question, "How tolerable was the cryocompression procedure for you?" on a scale from 0 to 100. A score of 0 means "not tolerable at all" and a score of 100 is "very tolerable". Pain, abnormal sensation, and adherence to cryocompression will also be evaluated as patient-reported measures of tolerability.
Acceptability: scale | Up to two months after completion of chemotherapy, an average of 6 months
  Subjects will be asked to complete a cryocompression acceptability assessment after each chemotherapy session in which they answer the questions, "How acceptable was the cryocompression procedure to you?" and "How likely are you to continue with cryocompression at your next chemotherapy treatment?" on a scale from 0 to 100, with 0 being "not acceptable, not likely to continue" and 100 being "very acceptable, very likely to continue".
Measure of manageability and acceptability for staff involved in the participants' care | Up to two months after completion of chemotherapy, an average of 6 months
  Staff will be asked to complete an acceptability assessment after each chemotherapy session in which they will answer the question, "How manageable or acceptable was this patient's cryotherapy/cryocompression therapy to you in working with a patient receiving chemotherapy?" on a scale from 0 to 100. A score of 0 means "not at all acceptable" and a score of 100 is "complete acceptable". They will also be asked "In your experience, compare the ease of use of the cryotherapy wrap versus plastic ice bags" on a scale from 0 to 100. A score of 0 means "cryotherapy wraps are much harder," and a score of 100 means "cryotherapy wraps are much easier."
Change in Patient Neurotoxicity Questionnaire [PNQ] (patient reported assessment) over time | Up to two months after completion of chemotherapy, an average of 6 months
  PNQ is a patient-reported questionnaire that consists of 2 items, representing motor and sensory components, with increasing grades for worsening symptoms. Patients will respond to each question for each of their 4 extremities by grading sensory and motor symptoms as A (no neuropathy), B (mild neuropathy), C (moderate neuropathy that does not interfere with activities of daily living [ADL]), D (moderate neuropathy that does interfere with ADL), or E (severe neuropathy that interferes with ADL).
Chemotherapy Dose | Up to two months after completion of chemotherapy, an average of 6 months
  Study staff will record the taxol dose at each cycle

CONTACTS AND LOCATIONS:
Overall Officials: Laura Havrilesky, Principal Investigator — DUHS
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Carilion Clinic, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No